CLINICAL TRIAL: NCT04490239
Title: Intranasal Heparin Tolerability Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua Sharp (Other)
Responsible Party: Sponsor-Investigator, Joshua Sharp, Associate Professor, University of Mississippi, Oxford
Organization: University of Mississippi, Oxford (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Intranasal Heparin
Record Dates: First submitted 2020-07-20; First posted 2020-07-29 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study will evaluate the acute and multi-day (14 days) tolerability of intranasally administered heparin. Two doses will be tested in the acute phase: 1000 U/day, then 2000 U/day. In the multi-day phase, the highest tolerated dose from the acute phase will be tested over a 14-day period of daily self-administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Subjects will be administered heparin sodium (porcine) bottled in a nasal sprayer with a volume per spray of 0.1 mL.
  Acute phase:
  On day 1, each subject will be administered 0.1 mL per nostril of 5000 U/mL heparin sodium (porcine), for a total dose of 1000 U. Vital signs, blood work, and follow-up clinical observation will be used to detect adverse effects.
  On day 2, each subject will be administered 0.1 mL per nostril of 10000 U/mL heparin sodium (porcine), for a total dose of 2000 U. Vital signs, blood work, and follow-up clinical observation will be used to detect adverse effects.
  Chronic phase:
  The highest acute dose that has no impact on aPTT or INR will be used for the chronic phase of this study. Each subject will be administered a daily dose for fourteen days. The first and last dose will be administered in the clinic; all other doses will be self-administered by subjects at home at the same time of day using a dosing diary to keep records.
  Interventions: Drug: Intranasal heparin sodium (porcine)

INTERVENTIONS:
Drug: Intranasal heparin sodium (porcine) — Intranasal heparin sodium
  Other Names: NDC (National Drug Code) 0409-2721-30; NDC 0409-2723-01

SUMMARY:
The investigators are investigating the tolerability of Heparin Sodium (porcine) administered topically via a nasal spray. This agent is being investigated as a potential prophylactic treatment to prevent infection by SARS(severe acute respiratory syndrome)-CoV-2, the novel coronavirus that causes COVID-19. Heparin Sodium (porcine) is an FDA-approved anticoagulant drug administered by injection. Recent work from multiple groups have found that heparin can prevent the infection of cells by SARS-CoV-2, indicating a possible use as a topical anti-viral. Numerous studies in both rodent models and humans have shown that heparin administered via a pulmonary or intranasal route enters the blood stream in negligible amounts, suggesting intranasal administration of heparin should be safe even at very large doses. Data from mouse models indicate that repeated daily nasal administration of heparin had no adverse effects in mice over a two week period (including weight loss, nose bleeds, loss of sense of smell, nasal discharge, or decreased blood clotting time). However, no data of repeated nasal administration of heparin in humans is available.

The investigators will test nasal administration of FDA-approved heparin sodium (porcine), originally formulated for injection. The formulations the investigators will be testing consist of heparin, sodium chloride, and 1% benzyl alcohol as a preservative bottled in a nasal sprayer dispensing 0.1 mL(millilitres) per spray. The investigation is planned in two phases. A single-dose phase will test the acute tolerability of the drug. In this phase, subjects will be administered 0.1 mL of Heparin Sodium in each nostril formulated at one of two doses: Day 1 will test a formulation of 5000 U(units)/mL, and Day 2 will test a formulation of 10000 U(units) /mL. After each dose, subjects will be tested for systemic exposure via blood aPTT tests and platelet count, as well as for local topical toxicity via examination for epistaxis and anosmia, along with any other adverse events. In the chronic phase, subjects will be administered the highest dose that was tolerated in the acute phase daily for fourteen days. Subjects will be tested for aPTT and platelet count, as well as epistaxis, anosmia and any other adverse events.

DETAILED DESCRIPTION:
Study Objectives

This exploratory clinical trial is designed to assess tolerability of increasing doses of intranasally administered heparin sodium in saline solution. Baseline values for aPTT and complete blood count will be obtained from six subjects. Heparin will be administered in increasing concentrations using one 0.1 mL(millilitre) spray per nostril (0.2 ml total) on a daily basis. Major signs of toxicity will be clinically relevant changes in aPTT time, clinically relevant decrease in platelet count, signs of anosmia 30 minutes after administration, or epistaxis. Dosing will start at 1000 units of heparin administered (500 units in each nostril) and then escalated to 2000 units. Should a clinically relevant aPTT prolongation (>50% increase from subject baseline) or decrease in platelet count (below clinical lab normal limit) be observed at either dose, the study will be halted and a series of lower doses evaluated.

Study Overview

Description of Design of Study

This study is a single center, prospective, Phase 0 exploratory tolerability trial. A total of 6 healthy subjects (3 M and 3 F) will be enrolled into the study. This study will evaluate the acute and multi-day (14 days) tolerability of intranasally administered heparin.

Test Article

Investigational Product

The study will assess the single and multi-dose tolerability of intranasal administration of an aliquot of an FDA-approved heparin sodium injection (5,000 USP units/mL or 10,000 USP units/mL) to deliver 1000U (units) or 2000U of heparin sodium. Doses will be prepared and administered as follows:

1000 U = (2 x 0.1 mL(milliliter) of 5000U(units)/mL or one spray of 500 U in each nostril) 2000 U = (2 x 0.1 mL of 10000U/mL or one spray of 1000 U in each nostril)

The test article will be administered by transferring (4 mL) of sterile heparin sodium injection (5,000 USP units/mL or 10,000 USP units/mL) at ambient room temperature into intranasal spray bottles, one for each individual subject.

The test article will be administered within 4 weeks of preparation, and the remainder discarded after study completion.

Supplier The test article (Heparin Sodium USP) will be obtained from appropriate commercial sources.

Safety Assessments

Safety assessments will be completed as part of this single and multi-dose, pharmacokinetic study. Safety will be assessed prior to test article administration and at 24 post dose, in the acute phase. For safety assessments during the chronic phase, safety assessments will be assessed prior to test article administration , day 14 and day 15-post study. Test subject will be called every three (3) days for updates and subjective reports (adverse events), during 14 day, daily dose phase. Subject safety will be assessed by monitoring adverse events, clinical laboratory tests, vital signs, and physical examinations.

Laboratory parameters will be evaluated during screening and daily, to include the following:

* Complete Blood Count (WBC, RBC(red blood cell count), Hematocrit, Hemoglobin, MCV (mean corpuscular volume), Platelet Count)
* PT(prothrombin time)/INR (international normalized ratio) Baseline and post study
* Serum/Urine hCG ( human chorionic gonadotropin)baseline and predose
* Activated Partial Thromboplastin Time (aPTT)

Clinical Adverse Events

Clinical Adverse Events will be monitored throughout the study. However, such events are not anticipated during this trial due to the low systemic exposure of the test article being administered. However, local side effects of intranasal heparin, such as epistaxis or nasal congestion may result.

For any abnormal lab values, test subjects will be evaluated for any sign and symptoms, and labs will be redrawn, until stabilized or returned to baseline. Subjects will be referred to the primary physician for any continued care required.

ELIGIBILITY:
Inclusion Criteria:

Normal, healthy adults aged 18 to 65 years

Exclusion Criteria:

* Allergy to Heparin
* Currently taking any prescription blood thinners or anti-coagulants, or currently taking any intranasal medication
* Known history of anemia, thrombocytopenia, or other blood disorder
* Autoimmune disorders
* Known history of Neurologic/Psychiatric disorders
* Report of an active infection
* Subject is pregnant or breast-feeding, or is expecting to conceive during the study.

NOTE: Subjects will be instructed to abstain from alcohol for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Gurley, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- The University of Mississippi National Center for Natural Products Research, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 36 months following publication
Access Criteria: Proposals should be directed to jsharp@olemiss.edu. To gain access, requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Tandon R, Sharp JS, Zhang F, Pomin VH, Ashpole NM, Mitra D, Jin W, Liu H, Sharma P, Linhardt RJ. Effective Inhibition of SARS-CoV-2 Entry by Heparin and Enoxaparin Derivatives. bioRxiv [Preprint]. 2020 Jul 28:2020.06.08.140236. doi: 10.1101/2020.06.08.140236. PMID 32577638

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Subjects will be administered heparin sodium (porcine) bottled in a nasal sprayer with a volume per spray of 0.1 mL.
  Acute phase:
  On day 1, each subject will be administered 0.1 mL per nostril of 5000 U/mL heparin sodium (porcine), for a total dose of 1000 U. Vital signs, blood work, and follow-up clinical observation will be used to detect adverse effects.
  On day 2, each subject will be administered 0.1 mL per nostril of 10000 U/mL heparin sodium (porcine), for a total dose of 2000 U. Vital signs, blood work, and follow-up clinical observation will be used to detect adverse effects.
  Chronic phase:
  The highest acute dose that has no impact on aPTT or INR will be used for the chronic phase of this study. Each subject will be administered a daily dose for fourteen days. The first and last dose will be administered in the clinic; all other doses will be self-administered by subjects at home at the same time of day using a dosing diary to keep records.
  Intranasal heparin sodium (porcine): Intranasal heparin sodium
Period: 1000 U Acute (One Dose, Day 1)
Arm/Group | Experimental Arm
Started | 6
Completed | 6
Not Completed | 0
Period: 2000 U Acute (One Dose, Day 3)
Arm/Group | Experimental Arm
Started | 6
Completed | 6
Not Completed | 0
Period: 2000 U Chronic (Daily, 14 Days)
Arm/Group | Experimental Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 31 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal or Abnormal Activated Partial Thromboplastin Time (aPTT), Acute Phase Day 1
Description: A measurement of blood clotting ability; tests for systemic bioavailability of intranasal heparin collected 24 hours after a 1000 U intranasal dose of heparin
Time Frame: 24 hours after a 1000 U intranasal dose of heparin
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Participants
  participants with normal aPTT (24-33 sec) | 6
  participants with abnormal aPTT (<24 sec or >33 sec) | 0

2. Primary Outcome: Number of Participants With Normal or Abnormal Activated Partial Thromboplastin Time (aPTT), Acute Phase Day 2
Description: A measurement of blood clotting ability; tests for systemic bioavailability of intranasal heparin collected 24 hours after a 2000 U intranasal dose of heparin
Time Frame: 24 hours after 2000 U dose intranasal heparin
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Participants
  Participants with normal aPTT (24-33 sec) | 6
  Participants with abnormal aPTT (<24 sec or >33 sec) | 0

3. Primary Outcome: Number of Participants With Normal or Abnormal Activated Partial Thromboplastin Time (aPTT), Chronic Phase Day 14
Description: A measurement of blood clotting ability; tests for systemic bioavailability of intranasal heparin obtained immediately after the 14 consecutive day of daily 2000 U dose of intranasal heparin
Time Frame: Day 14, chronic phase
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Participants
  Participants with normal aPTT (24-33 sec) | 6
  Participants with abnormal aPTT (<24 sec or >33 sec) | 0

4. Primary Outcome: Number of Participants With Normal or Abnormal Activated Partial Thromboplastin Time (aPTT), Chronic Phase Day 15
Description: A measurement of blood clotting ability; tests for systemic bioavailability of intranasal heparin obtained 24 hours after the 14 consecutive day of daily 2000 U dose of intranasal heparin
Time Frame: 24 hours after the last 2000 U dose of the chronic phase
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Participants
  Participants with normal aPTT (24-33 sec) | 6
  Participants with abnormal aPTT (<24 sec or >33 sec) | 0

5. Primary Outcome: Percent Change in Platelet Count From Pre-dose Baseline
Description: Indicative of heparin-induced thrombocytopenia, a serious adverse side effect of systemically bioavailable heparin, measured immediately after the last 2000 U intranasal dose of the chronic phase.
Time Frame: Pre-dose baseline, Day 14 chronic phase
Measure: Mean (Full Range); unit: percent change from baseline
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
percent change from baseline | 2.2 [-3.2 to 7.6]

6. Primary Outcome: Number of Incidents of Epistaxis, Acute Phase
Description: Number of incidents of blood coming from the nose during the acute phase
Time Frame: Day 0 through Day 2, acute phase
Measure: Number; unit: Reported incidents
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Reported incidents | 0

7. Primary Outcome: Number of Incidents of Epistaxis, Chronic Phase
Description: Blood coming from the nose or pink tinged nasal secretions
Time Frame: Day 1 through Day 15, chronic phase
Measure: Number; unit: Reported incidents
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Reported incidents | 1

8. Primary Outcome: Number of Participants With Normal or Abnormal Platelet Counts, Chronic Phase Day 14
Description: Abnormally low platelet counts indicative of heparin-induced thrombocytopenia, a serious adverse side effect of systemically bioavailable heparin, measured immediately after the last 2000 U intranasal dose of the chronic phase.
Time Frame: Day 14, Chronic Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Participants
  Participants with normal platelet counts (150,000 - 450,000 platelets/uL) | 6
  Participants with abnormal platelet counts (<150,000 or >450,000 platelets/uL) | 0

9. Secondary Outcome: Other Adverse Effects, Acute Phase
Description: Reports of mild, short-lived nasal irritation immediately after administration including mild burning sensation
Time Frame: Day 0 through Day 2, acute phase
Measure: Number; unit: Reported incidents
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Reported incidents | 2

10. Secondary Outcome: Other Adverse Effects, Chronic Phase
Description: Reports of mild, short-lived nasal irritation immediately after administration including mild burning sensation, itchiness or sneezing
Time Frame: Day 1 through Day 15, chronic phase
Measure: Number; unit: Reported incidents
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Reported incidents | 5

ADVERSE EVENTS:
Time Frame: From date of first dose in acute phase through sixteen days after last dose in chronic phase; 38 days total
Description: Adverse event collection was obtained by vital sign measurement, INR measurements from blood collection, and subject self-reporting
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=6)
Mild nasal irritation lasting less than 1 min after administration (Respiratory, thoracic and mediastinal disorders) | 2 (7) — Mild nasal irritation immediately after administration, lasting less than one minute. Includes mild burning sensation in the nose, itchiness and sneezing.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Incidents of mild nose bleeds and/or pink tinged nasal secretions (NOTE: affected subject disclosed prior history of epistaxis not initially disclosed during screening)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04490239/Prot_000.pdf